CLINICAL TRIAL: NCT02827292
Title: Effects of Peroperative Music on the Biomolecular Inflammatory Response In Laparoscopic Surgery: A Triple Blind Randomized Control Study
Brief Title: Effect of Music on Inflammatory Response During Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, PROF. BRIJ B AGARWAL, Vice Chairman, Department of Laparoscopic and General Surgery, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SirGangaRamH
Record Dates: First submitted 2016-05-05; First posted 2016-07-11 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Laparoscopy
Keywords: music; inflammation
MeSH Terms: conditions — Inflammation | interventions — Music Therapy; Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Surgery without music (Experimental): Intervention: Headphones without music (Silent). A headphone will be applied peroperatively but no music will be played. Blood samples to assess the biomolecular inflammatory response and the post operative monitoring will be done as per the protocol.
  Interventions: Other: No music; Procedure: Laparoscopic Surgery
- Laparoscopic Surgery with music (Experimental): Intervention: peroperative music via head phones. A headphone will be applied peroperatively and music will be played for the entire duration of the surgical procedure. Blood samples to assess the biomolecular inflammatory response and the post operative monitoring will be done as per the protocol.
  Interventions: Other: music; Procedure: Laparoscopic Surgery

INTERVENTIONS:
Other: music — A standard music with a standard volume as per the protocol will be played with headphones during the entire duration of the surgery starting from the point of induction to the time of extubation.
  A proper silent operative room environment will be maintained.
  Arms: Laparoscopic Surgery with music
Other: No music — Silent Headphones (Without music) will be applied to the patient from the point of induction of anaesthesia to the time of extubation.
  Arms: Laparoscopic Surgery without music
Procedure: Laparoscopic Surgery — Patients will undergo Laparoscopic Surgery as per the set protocol

SUMMARY:
This study evaluates the effect of per-operative music on the bio-molecular inflammatory response in laparoscopic surgery. Per-operative music intervention will be given to the test group via headphones while the control group will be applied headphones without any music (Silent). The inflammatory stress response will be measured postoperatively at 6 hours and 24 hours postoperatively along with the baseline levels measured preoperatively. The values will be compared between the test and control groups.

DETAILED DESCRIPTION:
Laparoscopic surgery (LS) has gained popularity both amongst surgeon as well as patients. The appeal of LS is based on improved patient reported outcomes (PRO). The main PROs like post operative pain, hospital stay and ability to return to activity are better with LS. The improvement in PROs has been attributed to attenuated post operative inflammatory response. The post operative inflammatory response has been studied by the changes in various cytokine pathways. The cytokine response has been shown to be subdued after LS as compare to conventional surgery. This benefit of subdued cytokine response has been shown to translate into better PROs.

Laparoscopic cholecystectomy (LC) has been considered an index LS. It is also an index LS for evaluation of potentially beneficial intervention in LS. The surgical discourse in last two decades has been to achieve clinical equivalence of LS with conventional surgery. The clinical outcomes with LC have stabilized. The current scientific discourse is geared towards improving PROs. A multi dimensional approach including pre-operative optimisation, protocoled anaesthesia technique, and 'systems approach' based surgery and standardised dissection techniques have been recommended.

Peri-operative music has been shown to improve PROs in LC . A recently published meta-analysis has established the benefits of peri-operative music in post operative convalescence. Peri-operative music has been shown to affect the neurohumoral and cyto-immune expressions of various 'cluster of differentiation' (CD) markers, on various cell lines.

Despite the established efficacy of music, there is reluctance amongst surgeon to adopt it routinely. There is no clarity and scientific curiosity about the type of music and the timing of music intervention, for the observed benefits of peri-operative music. The biomolecular basis of the reported benefits, of music in surgical setting has not been studied in an objective manner.

With this background the investigators hypothesized that per-operative music should have measurable bio-molecular footprint in postoperative convalescence use. With this hypothesis the investigators wish to study the per-operative music effects on the PROs, in laparoscopic cholecystectomy with measurable bio-molecular or/and bio-cellular markers.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years.
2. Should be able to understand and sign an informed consent.
3. Consent to the use of standard music during surgery.
4. Ability to maintain & communicate a PRO diary.
5. Ability to communicate via telephone or email or text message (SMS).
6. Fitness for general anaesthesia (ASA grade-I and ASA grade-II)

Exclusion Criteria:

1. Surgery for incidental Gall Bladder (GB) disease in patients for other surgeries.
2. Concomitant common bile duct (CBD) stone or any CBD intervention/pancreatitis in the preceding 6 weeks.
3. Non acceptance for the standard music or objection to any unknown music.
4. Suspicion of carcinoma gallbladder on ultrasonography
5. Patients with neuropathic pain/chronic pain needing regular anti-inflammatory drugs.
6. Documented or known sensitivity to any drug to be used in the study protocol.
7. Patient on immunosuppressant/ cytotoxic/ steroid therapy.
8. Pregnant or lactating ladies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Change in Interleukin 6 (IL-6) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of IL-6 will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery

SECONDARY OUTCOMES:
Change in Highly sensitive C-reactive protein (HS-CRP) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of HS-CRP will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in Tumor necrosis factor -α (TNF-α) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of TNF-α will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in CD-3+ (T cells) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of CD-3+ (T cells) will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in CD-3+/CD-4+ ratio | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of CD-3+/CD-4+ ratio will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in CD-3+/CD-8+ ratio | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of CD-3+/CD-8+ ratio will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in CD-19 (B cells) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of CD-19 (B cells) will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in Natural Killer Cells-(NK-Cells) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of NK-Cells will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery
Change in Immature platelet factor (IPF) | Baseline (preoperatively), 6hours postoperatively, 24 hours postoperatively
  serum levels of IPF will be measured preoperatively and postoperatively at 6 hours and 24 hours postoperatively to compare the inflammatory stress response to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Brij Bushan Agarwal, Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided